CLINICAL TRIAL: NCT05988450
Title: A Prospective, Multicenter, Single Arm Clinical Trial to Evaluate the Safety and Effectiveness of Transcatheter Mitral Valve Clip Delivery System and Steerable Guide Catheter in Patients With Moderate-severe or Severe Functional MR (FMR)
Brief Title: Safety and Effectiveness Study of SQ-Kyrin TMVr System for Functional Mitral Regurgitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVRP01-001A
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Functional Mitral Regurgitation
Keywords: Functional Mitral Regurgitation; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SQ-Kyrin TMVr System (Experimental): Transcatheter edge-to-edge mitral valve repair using SQ-Kyrin TMVr System.
  Interventions: Device: SQ-Kyrin Transcatheter Mitral Valve Repair System

INTERVENTIONS:
Device: SQ-Kyrin Transcatheter Mitral Valve Repair System — Transcatheter mitral valve clip placement to repair the valve and correct regurgitation.

SUMMARY:
To verify the safety and effectiveness of transcatheter mitral valve clip delivery system and steerable guide catheter produced by Shanghai Shenqi Medical Technology Co., Ltd. in patients with moderate-severe (3 +) or severe (4 +) functional MR (functional MR) who still have symptoms after full treatment.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single arm clinical study designed to evaluate the safety and effectiveness of transcatheter mitral valve clip delivery system and steerable guide catheter in patients with moderate-severe (3 +) or severe (4 +) functional MR (Functional MR) who still have symptoms after adequate treatment. This trial will be conducted at 41 sites in China and is planned to include a total of 118 subjects. All subjects received the trial device for transcatheter mitral valve clip delivery system and steerable guide catheter, and were followed up at 30 days, 6 months, and 12 months after surgery. The composite endpoint of all-cause death and hospitalization for heart failure was assessed at 12 months after surgery. After the 12th month follow-up, the statistical analysis, clinical summary and application for product registration were carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Severe functional MR (FMR) ≥3+ as determined by transthoracic echocardiography (TTE);
2. Note: Eligible TTE must be obtained at least 30 days after the subject has been stabilized on optimal therapy (including Guideline Directed Medical Therapy GDMT). In the judgment of the center's cardiac team, subjects have received adequate treatment according to applicable criteria, including treatment for coronary artery disease, left ventricular dysfunction, MR, and heart failure (e.g., with cardiac resynchronization therapy (CRT or CRT-D), implantable cardioverter-defibrillator (ICD) implantation, coronary revascularization, and stable GDMT (see Appendix III for the definition of GDMT).
3. Age ≥ 18 years old, regardless of gender;
4. Cardiac function classification NYHA class II, III or ambulatory IV a;
5. At least one hospitalization for heart failure or subjects with high BNP > 150 pg/ml or high NT-proBNP > 600 pg/ml in the past 12 months.
6. Note: BNP or NT-proBNP must be obtained after the subject has stabilized on optimal therapy including Guideline Directed Medical Therapy (GDMT) at least 30 days. The patients can understand the purpose of the trial, voluntarily participate and sign an informed consent form, and are willing to undergo relevant tests and clinical follow-up.
7. Left ventricular end-systolic diameter (LVESD)≤70mm
8. The MR beam mainly originates from the A2/P2 area
9. Mitral valve coaptation depth≤11mm, coaptation height≥2mm, effective length of anterior and posterior leaflets>10mm
10. Mitral valve effective orifice area (EOA) ≥ 4.0cm2

Exclusion Criteria:

1. History of mitral valve surgery;
2. Patients with infective endocarditis or suggestive of active infection;
3. Complicated with severe untreated coronary artery disease;
4. Patients with pulmonary hypertension (pulmonary systolic blood pressure>70mmHg);
5. patients with transthoracic echocardiographic evidence of moderate-severe to severe right ventricular dysfunction;
6. Left heart ejection fraction <20%;
7. Patients who are extremely frail and cannot tolerate general anesthesia surgery or is in the state of shock requiring circulatory support;
8. Patients diagnosed with hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis;
9. Severe renal insufficiency (eGFR ≤ 25 mL/min) or requiring chronic renal replacement therapy;
10. Patients with definite coagulation disorders and severe coagulation system diseases;
11. Patients with clear contraindications to the use of anticoagulants;
12. Patients with stroke or transient cerebral ischemic attack within 30 days;
13. Received cardiac pacemaker therapy or cardiac resynchronization therapy (CRT, CRT-D) or implanted cardioverter-defibrillator (ICD) implantation therapy within 30 days;
14. Any intracardiac mass, left ventricular or atrial thrombus detected on transthoracic echocardiography;
15. Severe tricuspid TR;
16. Patients with other valve disease requiring surgery or interventional therapy;
17. Patients with severe macrovascular disease requiring surgical treatment;
18. Severe symptomatic carotid stenosis (>70% on ultrasonography) or carotid stenting within 30 days;
19. Patients with inappropriate anatomical structures of the heart and valves indicated by imaging examinations;
20. Known allergy to contrast agents and nickel-titanium memory alloy products;
21. <Resting systolic blood pressure 90 mmHg or >160 mmHg;
22. Patients with diseases that seriously affect the evaluation of treatment, such as patients with severe neurological lesions affecting cognitive ability, patients with malignant tumors, etc.;
23. Patient life expectancy < 12 months;
24. Patients with severe thoracic deformity;
25. Women who are pregnant, breastfeeding, or planning to become pregnant within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause death and hospitalization for heart failure | 12 months
  Freefrom of all-cause death and hospitalization for heart failure

SECONDARY OUTCOMES:
Technical success rate | Immediate postoperative
  1. No surgical death
  2. Delivery system for successful delivery and retrieval of devices
  3. Successful devices release and accurate positioning
  4. No need for any emergency surgery related to the device or surgical approach
Device success rate | 30 days after surgery
  1. Successfully implanted valve clip
  2. Transthoracic echocardiographic assessment showing MR ≤2+
Surgical success rate | 30 days after surgery
  1. Device success
  2. No major adverse events occurred The major adverse event refers to the composite endpoint of death, stroke, myocardial infarction, and cardiovascular surgery due to device- or surgery-related adverse events following the atrial septum pathway via the femoral vein.
Rate of MR 2+ or less than 2+ at 30 days, 6 months, and 12 months after surgery; | 30 days, 6 months, and 12 months after surgery
  Rate of MR 2+ or less than 2+ at 30 days, 6 months, and 12 months after surgery;
Rate of hospitalization for heart failure at 30 days, 6 months, and 12 months after surgery; | 30 days, 6 months, and 12 months after surgery
  Rate of hospitalization for heart failure at 30 days, 6 months, and 12 months after surgery;
The rate of NYHA heart function class I or II at 30 days, 6 months, and 12 months after surgery; | 30 days, 6 months, and 12 months after surgery
  The rate of NYHA heart function class I or II at 30 days, 6 months, and 12 months after surgery;
Improvement in quality of life from baseline at 12 months after surgery (as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) score); | 12 months after surgery
  Improvement in quality of life from baseline at 12 months after surgery (as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) score);
Improvement in 6-minute walk distance from baseline at 12 months after surgery; | 12 months after surgery
  Improvement in 6-minute walk distance from baseline at 12 months after surgery;
Improvement in left ventricular end-diastolic volume (LVEDV) from baseline at 12 months after surgery; | 12 months after surgery
  Improvement in left ventricular end-diastolic volume (LVEDV) from baseline at 12 months after surgery;

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Ph.D, Principal Investigator — General Hospital of Northern Theater Command, PLA
Locations (1):
- General Hospital of Northern Theater Command, PLA, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu K, Zhu D, Jiang H, Chen J, Chen S, Zhang J, He B, Wang Y, Fu G, Chen J, An J, Xiu J, Guo X, Li Y, Cheng X, Li P, Chen Y, Zhou S, Sun Y, Yu B, Pan X, Han Y. One-Year Outcomes of Novel Transcatheter Edge-to-Edge Mitral Repair System in Patients With Functional Mitral Regurgitation. Catheter Cardiovasc Interv. 2025 Dec;106(7):3574-3582. doi: 10.1002/ccd.70230. Epub 2025 Oct 6. PMID 41054211